CLINICAL TRIAL: NCT00767260
Title: Autologous Bone Marrow Mononuclear Cell Infusion With Hyperbaric Oxygen Therapy in Type 2 Diabetes Mellitus
Brief Title: Bone Marrow Mononuclear Cell and Hyperbaric Oxygen Therapy in Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Principal Investigator, Jianming Tan, Vice President, Fuzhou General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: sc-dm-2008
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; bone marrow mononuclear cell; hyperbaric oxygen therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Health; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BM-MNC+HOT (Experimental): Autologous Bone Marrow Mononuclear cell Infusion Combined With Hyperbaric Oxygen Therapy
  Interventions: Drug: BM-MNC+HOT
- BM-MNC (Experimental): Autologous Bone Marrow mononuclear cell Infusion
  Interventions: Drug: BM-MNC
- HOT (Experimental): hyperbaric oxygen therapy
  Interventions: Device: HOT
- Control (Active Comparator): stand medical therapy (enhanced hemoglucose monitor, health and diet counseling and insulin injection)
  Interventions: Drug: SMT

INTERVENTIONS:
Drug: BM-MNC+HOT — Autologous Bone Marrow Mononuclear cell Infusion Combined With Hyperbaric Oxygen Therapy
  Arms: BM-MNC+HOT
Drug: BM-MNC — Autologous Bone Marrow Mononuclear cell Infusion
  Arms: BM-MNC
Device: HOT — Hyperbaric Oxygen Therapy
  Arms: HOT
Drug: SMT — hypoglycemic drugs or exogenous insulin
  Other Names: stand medical therapy (enhanced hemoglucose monitor, health and diet counseling and insulin injection)
  Arms: Control

SUMMARY:
There were evidences that the non-immune mediated inflammatory pathways of cell damage occurred in vitro in human islets upon hyperglycemia in type 2 diabetes mellitus. Autologous stem cell therapies were an emerging set of therapies that showed promise with a low side effect profile. we hypothesized that infusion of mononuclear cells from buffy coat obtained from bone marrow might provide multiple signals for regeneration and inflammation-induced lesion recovery of local tissues, of which the effect might be maximized by intra-arterial pancreatic infusion through angiography and combination with hyperbaric oxygen therapy.

This trail includes a foregoing sub-trial that investigate the feasibility and safety of a novel method for massive bone marrow collection. The traditional BM collecting procedure is unfavorable because it yields minor bone marrow. Studies have shown that physiological exercise can increase bone marrow blood flow, which might facilitate BM collection.

We plan to include a total of 60 patients with type 2 diabetes and randomly assign them to either a control group or an exercise group (n =30 each). The patients in the exercise group exercised 30 minutes before the operation. All patients underwent routine surgical care. The collected BM volume, operation time, collecting speed , puncture times and pain scores during the operation were recorded. Bone marrow samples were tested for CD34+ flow cytometry and whole blood cell count.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 40 to 65 years of age.
* Ability to provide written informed consent.
* Mentally stable and able to comply with the procedures of the study protocol.
* Clinical history compatible with type 2 diabetes (T2DM) as defined by the Expert Committee on the Diagnosis and classification of Diabetes Mellitus
* Onset of T2DM disease at ≥ 35 years of age.
* T2DM duration ≥ 3 and ≤ 20 years at the time of enrollment.
* Basal C-peptide 0.3-2.0 ng/mL
* HbA1c ≥ 7.5 and ≤ 12% before standard medical therapy (SMT). Patients must have been treated with SMT for minimum of 4 months prior to randomization. Insulin dose and metformin doses should be stable over the 3 months prior to randomization.
* HbA1c ≥ 7.5 and ≤ 9.5% at time of randomization.
* Total insulin daily dose (TDD) at time of randomization should not exceed 1.0 units/day/kg

Exclusion Criteria:

* BMI >35 kg/m2.
* Insulin requirements of > 100 U/day.
* HbA1c >9.5%. (at the time of randomization)
* C-reactive protein (hs-CRP) >3.00
* Uncontrolled blood Pressure: SBP >160 mmHg or DBP >100 mmHg at the time of randomization.
* Evidence of renal dysfunction, serum creatinine > 1.5 mg/dl (males) and 1.4 mg/dl (females).
* Proteinuria > 300 mg/day
* Evidence of cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in past 6 months.
* For female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study. For male participants: intent to procreate 3 months before or after the intervention or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable
* Active infection including hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB. Positive tests are acceptable only if associated with a history of previous vaccination in the absence of any sign of active infection. Positive tests are otherwise not acceptable, even in the absence of any active infection at the time of evaluation
* Known active alcohol or substance abuse including cigarette/cigar smoking
* Baseline Hgb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/L), neutropenia (<1,500/L), or thrombocytopenia (platelets <100,000/L).
* A history of Factor V deficiency or other coagulopathy defined by INR >1.5, PTT >40, PT >15.
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patients with an INR >1.5.
* Acute or chronic pancreatitis.
* Symptomatic peptic ulcer disease.
* Hyperlipidemia despite medical therapy (fasting LDL cholesterol >130 mg/dl, treated or untreated; and/or fasting triglycerides > 200 mg/dl).
* Receiving treatment for a medical condition requiring chronic use of systemic steroids.
* Symptomatic cholecystolithiasis.
* Use of any investigational agents within 4 weeks of enrollment.
* Admission to hospital for any reason in the 14 days prior to enrollment (signing consent).
* Presence of active proliferative diabetic retinopathy or macular edema
* Any malignancy
* Abnormal liver function >1.5 x ULN
* Abdominal aortic aneurysm
* History of cerebro-vascular accident
* Any patient with acute or subacute decompensation from diabetes
* Any acute or chronic infectious condition that in the criteria of the investigator would be a risk for the patient.
* Subjects with hypoproteinemia, cachexia or terminal states
* Subjects with history of anorexia/bulimia
* Subjects with respiratory insufficiency
* Subjects with a history of chronic sinusitis (sinusitis lasting more than 8 weeks in the past year) or recurrent acute sinusitis (sinusitis lasting more than 4 weeks more than four times in the past year.
* Any contraindication to hyperbaric oxygen treatment
* Subjects that are being treated with any medication that could interfere with the outcome of the study such as: Sulfonylureas, Thiazolidinediones and glucagon like peptide 1 (GLP-1) analogues (Exenatide, Byetta), Pramlintide (Amylin), Dipeptidyl-peptidase IV (DPP-IV) inhibitors (i.e. Sitagliptin, Januvia)
* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-03; Primary Completion 2012-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
area under the curve of c-peptide | 1 year

SECONDARY OUTCOMES:
The incidence and severity of adverse events related to the stem cell infusion procedure | 1 year
The incidence and severity of adverse events related to the hyperbaric oxygen therapy | 1 year
HbA1c | 1 year
exogenous insulin requirements | 1 year
fasting hemoglucose | 1 year
fasting c-peptide | 1 year
area under the curve of serum insulin | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan, professor, Principal Investigator — professor
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Wu Z, Luo F, Wu Z, Tao X, Zou X, Tan J. Preoperative exercise facilitates abundant bone marrow collection in patients with type 2 diabetes for mononuclear cell therapy. Cytotherapy. 2015 Apr;17(4):454-7. doi: 10.1016/j.jcyt.2014.11.007. Epub 2015 Jan 2. PMID 25559146
- [Derived] Wu Z, Cai J, Chen J, Huang L, Wu W, Luo F, Wu C, Liao L, Tan J. Autologous bone marrow mononuclear cell infusion and hyperbaric oxygen therapy in type 2 diabetes mellitus: an open-label, randomized controlled clinical trial. Cytotherapy. 2014 Feb;16(2):258-65. doi: 10.1016/j.jcyt.2013.10.004. Epub 2013 Nov 28. PMID 24290656